CLINICAL TRIAL: NCT00710554
Title: A Double Blind, Randomized, Placebo Controlled, Parallel Group Study of Sativex® in the Treatment of Subjects With Peripheral Neuropathic Pain, Associated With Allodynia
Brief Title: A Study of Sativex® for Pain Relief of Peripheral Neuropathic Pain, Associated With Allodynia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GWCL0405
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Pain; Peripheral Neuropathy
Keywords: Pain; Peripheral Neuropathy; Allodynia
MeSH Terms: conditions — Pain; Peripheral Nervous System Diseases; Hyperalgesia | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Experimental)
  Interventions: Drug: Sativex
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex — containing THC (27 mg/ml):CBD (25 mg/ml), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Maximum permitted dose was eight actuations in any three hour period and 24 actuations (THC 65 mg: CBD 60 mg) in 24 hours
  Other Names: GW-1000-02
  Arms: Sativex
Drug: Placebo — containing peppermint oil, 0.05% (v/v), quinoline yellow, 0.005% (w/v), sunset yellow, 0.0025% (w/v), in ethanol:propylene glycol (50:50) excipient.
  Other Names: GW-4001-01
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Sativex® compared with placebo in relieving peripheral neuropathic pain associated with allodynia.

DETAILED DESCRIPTION:
This was a 15 week (one week baseline and fourteen weeks treatment period), multicentre, double blind, randomised, placebo controlled, parallel group study to evaluate the efficacy of Sativex® in subjects with PNP, associated with allodynia. Subjects were screened to determine eligibility and completed a seven-day baseline period. Subjects then returned to the centre for assessment, randomisation and dose introduction. Visits occurred at the end of weeks two, six, ten and at the end of the study (treatment week 14) or earlier if they withdrew. A follow up visit occurred 28 days after completion or withdrawal. Subjects in this study were given the opportunity to be enrolled in an open label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent.
* Male or female, aged 18 years or above.
* Ability (in the investigators opinion) and willingness to comply with all study requirements.
* Diagnosed with PNP of at least six months duration and in who pain is not wholly relieved with their current therapy.
* Presence of mechanical allodynia within the territory of the affected nerve(s) which has been confirmed by either a positive response to stroking the allodynic area with a SENSELABTM Brush 05 or to force applied by a 5.07 gram Semmes-Weinstein monofilament.
* Had at least one of the following underlying conditions, which caused their peripheral neuropathic pain; post herpetic neuralgia, peripheral neuropathy, focal nerve lesion, radiculopathy or Complex Regional Pain Syndrome (CRPS) type 2.
* The daily diary 0-10 NRS pain scores on days B2 - B7 of the baseline period were completed and summed to at least 24.
* Stable dose of regular pain medication and non-pharmacological therapies (including TENS) for at least 14 days prior to the screening visit and willingness for these to be maintained throughout the study. Where subjects were taking a medication containing paracetamol further instructions were provided, refer to Section 9.4.7.
* In the opinion of the investigator the subject has received or was currently receiving the appropriate PNP treatments for their condition.
* Agreement for the responsible authorities (as applicable in individual countries), their primary care physician, and their consultant, if appropriate, to be notified of their participation in the study.

Exclusion Criteria:

* Concomitant pain thought by the investigator to be of a nature or severity to interfere with the subject's assessment of their PNP.
* Receiving a prohibited medication and were unwilling to stop or comply for the duration of the study.
* Had CRPS type 1, cancer related neuropathic pain or neuropathic pain resulted from diabetes mellitus.
* Has used either cannabis (either for recreational or medical purposes) or cannabis based medications within the last year and were unwilling to abstain for the duration for the study.
* History of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* Known or suspected history of alcohol or substance abuse.
* History of epilepsy or recurrent seizures.
* Known or suspected hypersensitivity to cannabinoids or any of the excipients of the study medication.
* Evidence of cardiomyopathy.
* Experienced myocardial infarction or clinically relevant cardiac dysfunction within the last 12 months or had a cardiac disorder that, in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction.
* QT interval; of > 450 ms (males) or > 470 ms (females) at Visit 1.
* Secondary or tertiary AV block or sinus bradycardia (HR <50bpm unless physiological) or sinus tachycardia (HR>110bpm) at Visit 1.
* Diastolic blood pressure of <50 mmHg or >105 mmHg in a sitting position at rest for 5 minutes prior to randomisation.
* Impaired renal function i.e., creatinine clearance is lower than 50ml/min at Visit 1 and is indicative of renal impairment.
* Significantly impaired hepatic function, at Visit 1, in the Investigator's opinion.
* Female subjects of child bearing potential and male subjects whose partner was of child bearing potential, unless were willing to ensure that they or their partner used effective contraception during the study and for three months thereafter.
* If female, were pregnant or lactating, or were planning pregnancy during the course of the study and for three months thereafter.
* Received an IMP within the 12 weeks before Visit 1.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, may influence the result of the study, or the subject's ability to participate in the study.
* Following a physical exam, the subject had any abnormalities that, in the opinion of the investigator, would prevent the subject from safely participating in the study.
* Intention to donate blood during the study.
* Intention to travel internationally during the study.
* Previous randomisation into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2005-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mick Serpell, MB ChB, FRCA, Principal Investigator — Pain Clinic Office
Locations (1):
- Pain Clinic Office, Gartnavel General Hospital,, Glasgow, West Lothain, United Kingdom

REFERENCES:
- [Result] Serpell M, Ratcliffe S, Hovorka J, Schofield M, Taylor L, Lauder H, Ehler E. A double-blind, randomized, placebo-controlled, parallel group study of THC/CBD spray in peripheral neuropathic pain treatment. Eur J Pain. 2014 Aug;18(7):999-1012. doi: 10.1002/j.1532-2149.2013.00445.x. Epub 2014 Jan 13. PMID 24420962

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex: Each actuation delivered 100 μl (THC 2.7 mg and CBD 2.5 mg) up to a maximum of 24 actuations in any 24 hour period.
- Placebo: Each 100 ul actuation delivered the excipients plus colorants, up to a maximum of 24 actuations in any 24 hour period.
Period: Overall Study
Arm/Group | Sativex | Placebo
Started | 128 | 118
Completed | 79 | 94
Not Completed | 49 | 24
Not completed — Adverse Event | 24 | 7
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Lost to Follow-up | 7 | 1
Not completed — Lack of Efficacy | 11 | 12
Not completed — Receiving radiotherapy - prostate cancer | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex | Placebo | Total
Number analyzed (Participants) | 128 | 118 | 246
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 88 | 179
  >=65 years | 37 | 30 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (14.38) | 57 (14.07) | 57.3 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 65 | 150
  Male | 43 | 53 | 96
Region of Enrollment [Number; unit: participants]
  United Kingdom | 74 | 72 | 146
  Belgium | 8 | 7 | 15
  Canada | 3 | 2 | 5
  Czech Republic | 35 | 32 | 67
  Romania | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Peripheral Neuropathic Pain on a 0-10 Numerical Rating Scale (NRS) Score at the End of Treatment (15 Weeks)
Description: The peripheral neuropathic pain NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your pain or average pain in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of pain. A negative value indicates an improvement in pain score from baseline.
Time Frame: Day 7 to Day 98
Population: The efficacy analyses were conducted on data from all subjects who were randomised, received at least one dose of study medication and yielded on-treatment efficacy data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 77 | 92
units on a scale | -1.36 (2.02) | -0.84 (1.86)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The model used for the analysis of the end of study value was an analysis of covariance (ANCOVA) with baseline value as a covariate and treatment group and centre group as main effect. Due to the low power of the test for interaction, the test was performed at the 10% significance level as a possible indicator of an interactive effect. The null hypothesis was one of no difference between treatments; Test type: Superiority or Other; p = 0.139, ANCOVA; estimated mean treatment difference = -0.34, 95% CI 2-sided [-0.79 to 0.11]

2. Secondary Outcome: Change From Baseline in Neuropathic Pain Scale Score at the End of Treatment (15 Weeks)
Description: The NPS score is 0-100 sum of 10 individual pain scores (0-10 NRS, 0= no pain to 10 = most pain imaginable). A negative change from baseline indicates an improvement in pain.
Time Frame: Day 7 to Day 98
Population: The primary population for the analysis of efficacy was the full analysis set, which included all randomised subjects who received at least one dose of test treatment and had on-treatment efficacy data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 78 | 93
units on a scale | -11.57 (16.15) | -7.19 (19.65)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change from baseline in mean Neuropathic Pain Scale score was compared between treatment groups and centres using ANCOVA. The model was to include treatment and centre group as factors and baseline mean usage as a covariate; Test type: Superiority or Other; p = 0.198, ANCOVA; Estimated mean treatment difference = -2.86, 95% CI 2-sided [-7.22 to 1.50]

3. Secondary Outcome: Change From Baseline in Sleep Quality 0-10 Numerical Rating Scale Scores at the End of Treatment (15 Weeks)
Description: The sleep disruption NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate how your pain disrupted your sleep last night?" where 0 = did not disrupt sleep and 10 = completely disrupted (unable to sleep at all). A negative value indicates an improvement in sleep disruption score from baseline.
Time Frame: Day 7 to Day 98
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 81 | 86
units on a scale | -2.0 (2.70) | -1.2 (2.38)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change from baseline score was compared between treatment groups and centres using ANCOVA. The model was to include treatment and centre group as factors and baseline mean usage as a covariate; Test type: Superiority or Other; p = 0.007, ANCOVA; Estimated mean treatment difference = -0.83, 95% CI 2-sided [-1.43 to -0.23]

4. Secondary Outcome: Change in Baseline Mean Dynamic Allodynia Test Score at the End of Treatment (15 Weeks)
Description: Dynamic allodynia was assessed by stroking the skin over the affected area five times with a standardised brush, designed specifically for sensory testing at 5 s intervals, and recording the pain severity on a 0-10 point scale (0= no pain to 10 = most pain imaginable). All strokes were of the same length, minimum 2 cm. Each dynamic allodynia score was calculated as the average of the five strokes.A negative change from baseline indicates an improvement in score.
Time Frame: Day 7 and Day 98
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 112 | 102
units on a scale | -1.1 (2.16) | -1.0 (2.49)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in the dynamic allodynia pain score from baseline to the end of treatment was analysed using ANCOVA with the baseline value as a covariate and country and treatment group as factors; Test type: Superiority or Other; p = 0.795, ANCOVA; Estimated mean treatment difference = 0.08, 95% CI 2-sided [-0.52 to 0.68]

5. Secondary Outcome: Change in Baseline Mean Punctate Allodynia Test Scores at the End of Treatment (15 Weeks)
Description: Punctate allodynia was measured using an in-house built pressure algometer comprising a strain gauge connected to a metal filament with a diameter of 1 mm and blunt tip at baseline and end of study. The filament was manually directed against the skin at an angle of 90 degrees and a steadily increasing pressure applied until the patient verbally indicated that they perceived pain (punctate pressure pain threshold). Patients were asked to verbally rate the intensity of the pain elicited, choosing a number between 0 (no pain)and 10 (most intense pain imaginable).
Time Frame: Day 7 and Day 98
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 112 | 106
units on a scale | 0.2 (0.78) | 0.3 (1.08)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in the punctate allodynia pain threshold force from baseline to the end of treatment was analysed using ANCOVA with the baseline value as a covariate and country and treatment group as factors; Test type: Superiority or Other; p = 0.233, ANCOVA; Estimated mean treatment difference = -0.14, 95% CI 2-sided [-0.37 to 0.09]

6. Secondary Outcome: Subject Global Impression of Change
Description: A 7-point Likert-type scale was used, with the question: 'Please assess the status of your pain due to peripheral neuropathy since entry into the study using the scale below' with the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse or very much worse". At Visit 2 (Baseline) patients wrote a brief description of their pain caused by peripheral neuropathy which was used at end of treatment to aid their memory regarding their symptoms at study start. For each of above markers the number of participants were reported.
Time Frame: Day 98
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 117 | 111
participants
  Very much improved | 8 | 4
  Much improved | 16 | 10
  Slightly improved | 38 | 24
  No change | 44 | 66
  Slightly worse | 9 | 4
  Much worse | 2 | 3
Statistical Analysis 1: Comparison: Sativex vs Placebo; The two treatment groups were compared using ordinal logistic regression and the proportional odds model. The initial model incorporated treatment and centre group as factors. The odds ratio together with its 95% CI and associated p-value are presented; Test type: Superiority or Other; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 1.762, 95% CI 2-sided [1.08 to 2.88]

7. Secondary Outcome: Change From Baseline in Brief Pain Inventory (Short Form) Scores at the End of Treatment
Description: The BPI-SF is a 14-item questionnaire that asks patients to rate pain over the prior week and the degree to which it interferes with activities on a 0 to 10 scale, where 0=no pain and 10=pain as bad as you can imagine. Severity is measured as worst pain, least pain, average pain, and pain right now. The severity composite score was calculated as the arithmetic mean of the four severity items(range 0-10). The minimum value is zero and maximum is 10. A higher score represents a poor outcome.
Time Frame: Day 7 and Day 98
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 114 | 105
units on a scale | -0.9 (1.69) | -0.6 (1.90)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change from baseline in mean Brief Pain Inventory (short form) score was compared between treatment groups and centres using ANCOVA. The model was to include treatment and centre group as factors and baseline mean usage as a covariate; Test type: Superiority or Other; p = 0.288, ANCOVA; Estimated mean treatment difference = -0.25, 95% CI 2-sided [-0.72 to 0.21]

8. Secondary Outcome: Change From Baseline in Quality of Life EuroQol 5-D (Health Status Index) Score at the End of Treatment (15 Weeks)
Description: The EQ-5D questionnaire provided two outcomes:(1)A weighted health state index visual analogue scale (VAS); (2) A self-rated health status VAS. EQ-5D Health Status VAS Scale: 0 = worst health state imaginable to 100 = best health state imaginable. An increase in score indicates an improvement in condition.The weighted health state index used the same VAS as above but was calculated for each assessment without imputation to account for missing values i.e., if one or more individual items was missing then the whole index was missing.
Time Frame: Day 7 and Day 98
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 113 | 107
units on a scale | 0.037 (0.187) | 0.044 (0.214)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change from baseline in mean EuroQol-5D score was compared between treatment groups and centres using ANCOVA. The model included treatment and centre groups as factors and baseline mean usage as a covariate; Test type: Superiority or Other; p = 0.617, ANCOVA; Estimated mean treatment difference = -0.01, 95% CI 2-sided [-0.06 to 0.04]

9. Secondary Outcome: Change From Baseline in Quality of Life EuroQol 5-D (Health Status Visual Analogue Scale) Score at the End of Treatment (15 Weeks)
Description: The EQ-5D questionnaire provided two outcomes:(1)A weighted health state index visual analogue scale (VAS); (2) A self-rated health status VAS. EQ-5D Health Status VAS Scale: 0 = worst health state imaginable to 100 = best health state imaginable. An increase in score indicates an improvement in condition.
Time Frame: Day 7 and Day 98
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 111 | 105
units on a scale | 3.7 (20.6) | 2.5 (21.2)
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.76, ANCOVA; Median Difference (Final Values) = -0.75, 95% CI 2-sided [-5.60 to 4.09], Standard Error of Mean 2.459

10. Secondary Outcome: Change From Baseline in the Use of Rescue Analgesia at the End Treatment (15 Weeks)
Description: Use of break through medication was recorded daily during the study as the number of paracetamol tablets taken. The change in mean daily quantities of tablets used was calculated from baseline to the last seven days of treatment.
Time Frame: Days 0-7 and Days 92-98
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of tablets
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 77 | 92
number of tablets | -0.99 (2.20) | -0.47 (2.08)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The model used for the analysis of the end of study value was an ANCOVA with baseline value as a covariate and treatment group and centre group as main effect. The null hypothesis was one of no difference between treatments; Test type: Superiority or Other; p = 0.112, ANCOVA; Estimated mean treatment difference = -0.38, 95% CI 2-sided [-0.85 to 0.09]

11. Secondary Outcome: Incidence of Adverse Events as a Measure of Subject's Safety.
Description: The number of subjects that reported an adverse event in this study is presented.
Time Frame: 19 weeks
Population: All subjects were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 128 | 118
participants | 109 | 83

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the time of consent to post study follow up i.e. 19 weeks were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex | Placebo
Serious Adverse Events (participants affected / at risk) | 10/128 | 6/118
Other Adverse Events (participants affected / at risk) | 109/128 | 83/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=128) | Placebo (N=118)
Bronchopneumonia (Infections and infestations) | 1 | 0
Infective Exacerbation of Chronic Obstructive Airway Disease (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1
Breast Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Enterovesical Fistula (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Lumbar Vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=128) | Placebo (N=118)
Dizziness (Nervous system disorders) | 52 | 12
Dysgeusia (Nervous system disorders) | 14 | 2
Headache (Nervous system disorders) | 13 | 9
Disturbance in Attention (Nervous system disorders) | 8 | 2
Neuropathy Peripheral (Nervous system disorders) | 6 | 4
Tremor (Nervous system disorders) | 6 | 0
Somnolence (Nervous system disorders) | 5 | 2
Balance Disorder (Nervous system disorders) | 4 | 2
Memory Impairment (Nervous system disorders) | 4 | 2
Sedation (Nervous system disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 23 | 14
Vomiting (Gastrointestinal disorders) | 13 | 7
Diarrhoea (Gastrointestinal disorders) | 12 | 6
Dry Mouth (Gastrointestinal disorders) | 11 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 6 | 4
Constipation (Gastrointestinal disorders) | 4 | 2
Mouth Ulceration (Gastrointestinal disorders) | 4 | 6
Oral Pain (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 20 | 8
Feeling Drunk (General disorders) | 8 | 3
Application Site Pain (General disorders) | 7 | 2
Dissociation (Psychiatric disorders) | 9 | 0
Disorientation (Psychiatric disorders) | 8 | 0
Depression (Psychiatric disorders) | 6 | 0
Anxiety (Psychiatric disorders) | 4 | 1
Panic Attack (Psychiatric disorders) | 4 | 1
Nasopharyngitis (Infections and infestations) | 9 | 8
Gastroenteritis (Infections and infestations) | 4 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 4 | 3
Increased Appetite (Metabolism and nutrition disorders) | 6 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 4
Vertigo (Ear and labyrinth disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.